CLINICAL TRIAL: NCT03769493
Title: Mobile After-Care Support Intervention for Patients With Schizophrenia Following Hospitalization (MACS)
Brief Title: Mobile After-Care Intervention to Support Post-Hospital Transition (MACS)
Acronym: MACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Brandon Gaudiano, Research Psychologist, Butler Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1806-001; R34MH115144 (NIH)
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Psychotic Disorders
Keywords: Medication adherence; Treatment adherence; Ecological momentary assessment; Ecological momentary intervention; Coping skills; Psychiatric Hospitalization
MeSH Terms: conditions — Psychotic Disorders; Medication Adherence; Treatment Adherence and Compliance | interventions — Amyloid

STUDY DESIGN:
Intervention Model Description: An uncontrolled open trial approach will be used in which all participants receive the MACS app.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile After-Care Support (MACS) app (Experimental): All participants will download the MACS app to their mobile phone (or a study provided phone, as needed). The app runs through the third-party platform, mEMA, designed by Ilumivu. It is designed to prompt engagement through questions and tailored responses at multiple times throughout the day and provide brief interventions.
  Interventions: Behavioral: Mobile After-Care Support (MACS) app

INTERVENTIONS:
Behavioral: Mobile After-Care Support (MACS) app — The MACS app assesses and intervenes by fostering increased treatment adherence (medication/appointments) and self-coping with illness (active, planned, problem-solving focused) to reduce symptoms and improve functioning. Additionally, MACS encourages participants who are already reporting adherence and healthy coping by using positive reinforcement strategies to maintain efforts and promote additional goal setting. MACS app strategies are linked to participants' specific assessment responses, allowing for a highly personalized self-management intervention experience. The MACS app provides interactive exercises delivered by the device designed to teach patients coping skills that they can use now and in the future.

SUMMARY:
This study examines the feasibility and acceptability of a mobile device-delivered app, called Mobile After-Care Support (MACS), to improve patients' coping and treatment adherence following a hospitalization related to their psychotic-spectrum disorder.

DETAILED DESCRIPTION:
In the open trial, all participants will receive a study-developed app to be used on a mobile phone. This app will support the use of healthy coping skills post-hospitalization, as well as help participants adhere to their discharge treatment plan. This phase is intended to inform the feasibility and acceptability of the app in preparation for a future randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Currently hospitalized
2. DSM-5 criteria for psychotic disorder (schizophrenia or schizoaffective disorder)
3. 18 years or older
4. Prescribed oral antipsychotic medication upon discharge
5. Ability to speak and read English

Exclusion Criteria:

1. Alcohol/drug use disorders at moderate or severe level
2. Planned discharge to supervised living setting or participation in formal outpatient adherence programs (e.g., medication packaging)
3. Pregnancy or other medical condition (e.g., dementia) contraindicating use of antipsychotic medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon A Gaudiano, Ph.D., Principal Investigator — Butler Hospital & Brown Universit; Ethan Moitra, Ph.D., Principal Investigator — Brown University
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Data available on the National Institute of Mental Health Data Archive (NDA).
Time Frame: Currently available.
Access Criteria: See NDA web site for details.
URL: https://nda.nih.gov/

REFERENCES:
- [Result] Moitra E, Park HS, Gaudiano BA. Development and Initial Testing of an mHealth Transitions of Care Intervention for Adults with Schizophrenia-Spectrum Disorders Immediately Following a Psychiatric Hospitalization. Psychiatr Q. 2021 Mar;92(1):259-272. doi: 10.1007/s11126-020-09792-9. PMID 32613525
- See also: Development and initial testing of an mHealth transitions of care intervention for adults with schizophrenia-spectrum disorders immediately following a psychiatric hospitalization — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7775867/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile After-Care Support (MACS) App
Started | 10
Completed | 7
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Mobile After-Care Support (MACS) App
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction Questionnaire (CSQ)
Description: The Client Satisfaction Questionnaire is a self-report measure of patient satisfaction with treatment. The total score will be used and ranges from 8 to 32 with increased scores indicating greater satisfaction with treatment.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mobile After-Care Support (MACS) App
Number analyzed (Participants) | 7
units on a scale | 19.2 (1.6)

2. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS)
Description: The interviewer-rated BPRS is a measure of psychiatric symptom severity. The total score will be used to assess overall severity with scores ranging from 18 to 126 and higher scores indicating greater severity.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile After-Care Support (MACS) App
Number analyzed (Participants) | 7
score on a scale
  Baseline | 46.4 (6.7)
  1 Month | 30.4 (8.5)
Statistical Analysis 1: Comparison: Mobile After-Care Support (MACS) App; Test type: Superiority; p < .001, t-test, 2 sided

3. Secondary Outcome: Brief Adherence Rating Scale (BARS)
Description: The BARS assesses the percentage of missed medication doses over the past month. The total adherence score ranges from 0% to 100% and higher scores indicate greater adherence.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile After-Care Support (MACS) App
Number analyzed (Participants) | 7
score on a scale
  Baseline | 96.7 (8.8)
  1 Month | 97.5 (4.6)
Statistical Analysis 1: Comparison: Mobile After-Care Support (MACS) App; Test type: Superiority; p = .875, t-test, 2 sided

4. Secondary Outcome: Maastricht Assessment of Coping Strategies (MACS)
Description: The MACS is an interviewer-rated assessment of the coping strategies that patients report using to manage their symptoms.
Time Frame: 1 month
Population: No data were collected for this measure (MACS). This is because we were unable to administer the measure as originally planned.
Arm/Group | Mobile After-Care Support (MACS) App
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Mobile After-Care Support (MACS) App
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mobile After-Care Support (MACS) App (N=10)
Rehospitalization (Psychiatric disorders) | 1

LIMITATIONS AND CAVEATS:
This is a treatment development study and therefore was not designed to test the efficacy of the intervention given the small sample size. Instead, the goal was examine feasibility and acceptability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT03769493/Prot_SAP_000.pdf